CLINICAL TRIAL: NCT05726734
Title: Efficacy of Vonoprazan-containing Triple Therapy Versus Empiric Bismuth Quadruple Therapy for First-line Helicobacter Pylori Treatment: a Randomized Clinical Trial
Brief Title: Vonoprazan-containing Triple Therapy Versus Empiric Bismuth Quadruple Therapy for First-line Helicobacter Pylori Treatment: a Randomized Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Principal Investigator, Yingjie Ji, Medical Doctor of Division of Endoscopy Center, Department of Gastroenterology of Shanghai East Hospital, Shanghai East Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022150
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori Infection
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Metronidazole; Esomeprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan-containing Triple Therapy (Active Comparator): Vonoprazan 20mg bid, Amoxicillin 1.0g tid and Metronidazole 0.4g tid for 14 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin, Metronidazole
- Empiric Bismuth Quadruple Therapy (Experimental): Esomeprazole 20mg bid, Bismuth Potassium Citrate 600mg bid, Amoxicillin 1.0g tid and Metronidazole 0.4g tid for 14 days
  Interventions: Drug: Amoxicillin, Metronidazole; Drug: Bismuth Potassium Citrate; Drug: Esomeprazole

INTERVENTIONS:
Drug: Vonoprazan — potassium-competitive acid blocker
  Arms: Vonoprazan-containing Triple Therapy
Drug: Amoxicillin, Metronidazole — Antibiotics for H. pylori eradication
Drug: Bismuth Potassium Citrate — Gastric mucosal protective drug with anti-H. pylori effect
  Arms: Empiric Bismuth Quadruple Therapy
Drug: Esomeprazole — Proton pump inhibitor
  Arms: Empiric Bismuth Quadruple Therapy

SUMMARY:
Vonoprazan Amoxicillin and metronidazole based triple therapy had achieved a high cure rate in the rescue treatment of helicobacter pylori infection. This study aims to evaluate the efficacy and safety of the Vonoprazan, amoxicillin and metronidazole based triple therapy and the empiric bismuth quadruple therapy in the naive patients with Helicobacter pylori infection.

ELIGIBILITY:
Inclusion Criteria:

* Participants with non-ulcer functional dyspepsia or peptic ulcer disease
* Ability and willingness to participate in the study and to sign and give informed consent
* Confirmed H. pylori infection and with no previous treatment experience

Exclusion Criteria:

* Less than 18 years old
* With previous gastric surgery
* Major systemic diseases
* Pregnancy or lactation
* Allergy to any of the study drugs Administration of antibiotics, bismuth, antisecretory drugs in 8 weeks prior to inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-06 (Estimated); Primary Completion 2025-02-06 (Estimated); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | Six weeks after completion of therapy
  Six weeks after completion of therapy, H. pylori eradication was assessed by ¹³C-urea breath test. Eradication was defined as negative result from urea breath test (<4‰) (4‰ as the cutoff value).

SECONDARY OUTCOMES:
Rate of adverse effects | Within 7 days after completion of therapy
  The subjects were asked to grade the severity of adverse events according to their influence on daily activities, experienced as "mild" (transient and well tolerated), "moderate" (causing discomfort and partially interfering with daily activities), or "severe" (causing considerable interference with daily activities)
Compliance rate | Within 7 days after completion of therapy
  Compliance was defined as poor when they had taken less than 80% of the total medication

CONTACTS AND LOCATIONS:
Overall Officials: Yingjie Ji, M.D., Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No